CLINICAL TRIAL: NCT01498601
Title: Improving Oral Care to Reduce Hospital Acquired Pneumonia (HAP) in the Acute, Non-Intubated, Care Dependent, Neurologically Impaired Adult Patient Population
Brief Title: Improving Oral Care to Reduce Hospital-Acquired Pneumonia (HAP) in the Acute Neurologically Impaired Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDAAA
Record Dates: First submitted 2011-12-13; First posted 2011-12-23 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2011-12

CONDITIONS: Pneumonia
Keywords: oral hygiene; tracheostomy; deglutition disorders; enteral nutrition; brain injury; coma
MeSH Terms: conditions — Pneumonia; Deglutition Disorders; Brain Injuries; Coma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral care treatment group (Experimental): All subjects in the prospective intervention group will receive the same enhanced oral care protocol
  Interventions: Other: Enhanced oral care protocol
- Retrospective study group (No Intervention): For comparison purposes, a retrospective chart review of matched in-patient population will reveal pneumonia rates in the same population who did not receive the enhanced oral care protocol.

INTERVENTIONS:
Other: Enhanced oral care protocol — * Changing mouth suction equipment every 24 hours
  * Mouth assessment every 2-4 hours
  * Cleansing mouth with toothbrush every 12 hours
  * Cleansing oral mucosa with oral rinse solution every 2-4 hours
  * Moisturize mouth/lips with swab and standard mouth moisturizer every 4 hours
  * Suction mouth and throat as needed
  * Head of the bed elevated to a minimum of 30° during oral care
  Other Names: Sage oral care products
  Arms: Oral care treatment group

SUMMARY:
Hypothesis: The investigators hypothesize that the current oral protocol is sub-optimal and an enhanced protocol will decrease the incidence of hospital acquired pneumonia (HAP)in the acute, non-intubated, care-dependent, neurologically impaired, adult patient.

DETAILED DESCRIPTION:
Overview Problem: Hospital-acquired pneumonia (HAP) is the second most common nosocomial infection and is a significant cause of morbidity and mortality. In the surgical population, HAP is associated with a 55% increase in length of stay and increased costs of approximately $31,000.00 per case. Neurologically impaired patients (those with brain injury causing alterations in mental status, immobility, impaired swallowing and cough, and increased risk of aspiration) are particularly vulnerable to HAP. HAP negatively impacts patient comfort and satisfaction, increases costs associated with diagnostic tests and treatments, increases risk for sepsis, and potential for higher level of care. It is estimated 95% of care-dependent patients on the Royal Columbian Hospital (RCH) neuroscience unit acquire HAP during their stay.

Gap: Research studies have shown improving oral hygiene in critical care, neuroscience intensive care units and cardiac surgery reduces the incidence of HAP. However, in the acutely ill neuroscience population outside critical care areas, this relationship has not been determined. Current oral care protocols, products and practitioner practice on medical/surgical units such as the RCH neuroscience unit do not consider recent evidence or recent increases in patient acuity and complexity.

Goal: The goal of this study is to test the efficacy of an improved, evidence-based oral care protocol in reducing HAP in this population on the medical/surgical neuroscience unit at RCH.

Research question: Does implementing an enhanced oral care protocol reduce rates of HAP in the acute, non-intubated, care-dependent, neurologically impaired, adult patient on a neuroscience unit?

Objective: To measure and compare the incidence of HAP among medical/surgical patients who had the current standard of oral care with those receiving an improved, preventative-based, oral hygiene protocol including regular teeth brushing, mouth and tongue inspection, swabbing and moisturizing, elevation of head of the bed (HOB), changing of suction equipment, and universal precautions.

Relevance: This study may identify the importance of standardizing oral hygiene protocols to the evidence, and heighten awareness among care providers in the prevention of HAP. If proven successful, the oral care protocol could be considered for implementation on acute units outside the RCH neuro unit.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 19 years)
* Admitted to RCH neuroscience unit
* Primary diagnosis is neurological (brain injury/insult)
* Non-intubated
* Dependent for oral care and unable to direct their own oral care

Exclusion Criteria:

* < 19 years
* Off service patients
* Intubated, on bilevel positive airway pressure or continuous positive airway pressure devices, (respiratory assistive devices)
* Palliative
* Capable of directing their own oral care
* Unable to receive oral care due to: oral tubes, nasal/oral airways, wired jaws, or behaviours such as resistiveness, combativeness, non-compliance, etc.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trudy L. Robertson, MSN, Principal Investigator — Fraser Health Authority; Dulcie J. Carter, MMedSci, Principal Investigator — Fraser Health Authority
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

REFERENCES:
- [Background] Marik PE. Aspiration pneumonitis and aspiration pneumonia. N Engl J Med. 2001 Mar 1;344(9):665-71. doi: 10.1056/NEJM200103013440908. No abstract available. PMID 11228282
- [Background] Marik PE, Kaplan D. Aspiration pneumonia and dysphagia in the elderly. Chest. 2003 Jul;124(1):328-36. doi: 10.1378/chest.124.1.328. PMID 12853541
- [Background] Munro CL, Grap MJ. Oral health and care in the intensive care unit: state of the science. Am J Crit Care. 2004 Jan;13(1):25-33; discussion 34. PMID 14735645
- [Background] Perry & Potter. Fraser Health Nursing Skills for Mouth Care for the Unconscious or Debilitated Patient. Mosby's Nursing Skills: Clinical Nursing Skills & Techniques (7th Ed.). St. Louis. Retrieved April 14th, 2011 from: http://app44.webinservice.com/NursingSkills/ContentPlayer/SkillContentPlayerIFrame.aspx?KeyId=598&Id=GN_14_3&Section=1&bcp=Index~M~False&IsConnect=False
- [Background] Shigemitsu H, Afshar K. Aspiration pneumonias: under-diagnosed and under-treated. Curr Opin Pulm Med. 2007 May;13(3):192-8. doi: 10.1097/MCP.0b013e3280f629f0. PMID 17414126
- [Background] Terpenning MS, Taylor GW, Lopatin DE, Kerr CK, Dominguez BL, Loesche WJ. Aspiration pneumonia: dental and oral risk factors in an older veteran population. J Am Geriatr Soc. 2001 May;49(5):557-63. doi: 10.1046/j.1532-5415.2001.49113.x. PMID 11380747
- [Result] American Association of Critical Care Nurses. AACN Practice Alert: Oral Care for Patients at Risk for Ventilator-Associated Pneumonia. Retrieved April 10, 2011 from: http://www.aacn.org
- [Result] Bopp M, Darby M, Loftin KC, Broscious S. Effects of daily oral care with 0.12% chlorhexidine gluconate and a standard oral care protocol on the development of nosocomial pneumonia in intubated patients: a pilot study. J Dent Hyg. 2006 Summer;80(3):9. Epub 2006 Jul 1. PMID 16953990
- [Result] Chan EY, Ruest A, Meade MO, Cook DJ. Oral decontamination for prevention of pneumonia in mechanically ventilated adults: systematic review and meta-analysis. BMJ. 2007 Apr 28;334(7599):889. doi: 10.1136/bmj.39136.528160.BE. Epub 2007 Mar 26. PMID 17387118
- [Result] Cohn JL, Fulton JS. Nursing staff perspectives on oral care for neuroscience patients. J Neurosci Nurs. 2006 Feb;38(1):22-30. doi: 10.1097/01376517-200602000-00006. PMID 16568810
- [Result] DeRiso AJ 2nd, Ladowski JS, Dillon TA, Justice JW, Peterson AC. Chlorhexidine gluconate 0.12% oral rinse reduces the incidence of total nosocomial respiratory infection and nonprophylactic systemic antibiotic use in patients undergoing heart surgery. Chest. 1996 Jun;109(6):1556-61. doi: 10.1378/chest.109.6.1556. PMID 8769511
- [Result] Fields LB. Oral care intervention to reduce incidence of ventilator-associated pneumonia in the neurologic intensive care unit. J Neurosci Nurs. 2008 Oct;40(5):291-8. doi: 10.1097/01376517-200810000-00007. PMID 18856250
- [Result] Grap MJ, Munro CL, Ashtiani B, Bryant S. Oral care interventions in critical care: frequency and documentation. Am J Crit Care. 2003 Mar;12(2):113-8; discussion 119. PMID 12625169
- [Result] Hilker R, Poetter C, Findeisen N, Sobesky J, Jacobs A, Neveling M, Heiss WD. Nosocomial pneumonia after acute stroke: implications for neurological intensive care medicine. Stroke. 2003 Apr;34(4):975-81. doi: 10.1161/01.STR.0000063373.70993.CD. Epub 2003 Mar 13. PMID 12637700
- [Result] Houston S, Hougland P, Anderson JJ, LaRocco M, Kennedy V, Gentry LO. Effectiveness of 0.12% chlorhexidine gluconate oral rinse in reducing prevalence of nosocomial pneumonia in patients undergoing heart surgery. Am J Crit Care. 2002 Nov;11(6):567-70. PMID 12425407
- [Result] Langmore SE, Terpenning MS, Schork A, Chen Y, Murray JT, Lopatin D, Loesche WJ. Predictors of aspiration pneumonia: how important is dysphagia? Dysphagia. 1998 Spring;13(2):69-81. doi: 10.1007/PL00009559. PMID 9513300
- [Result] Prendergast V, Hallberg IR, Jahnke H, Kleiman C, Hagell P. Oral health, ventilator-associated pneumonia, and intracranial pressure in intubated patients in a neuroscience intensive care unit. Am J Crit Care. 2009 Jul;18(4):368-76. doi: 10.4037/ajcc2009621. PMID 19556415
- [Result] Reimer-Kent J. From theory to practice: preventing pain after cardiac surgery. Am J Crit Care. 2003 Mar;12(2):136-43. PMID 12625171
- [Result] Rotstein C, Evans G, Born A, Grossman R, Light RB, Magder S, McTaggart B, Weiss K, Zhanel GG. Clinical practice guidelines for hospital-acquired pneumonia and ventilator-associated pneumonia in adults. Can J Infect Dis Med Microbiol. 2008 Jan;19(1):19-53. doi: 10.1155/2008/593289. PMID 19145262
- [Result] Safdar N, Crnich CJ, Maki DG. The pathogenesis of ventilator-associated pneumonia: its relevance to developing effective strategies for prevention. Respir Care. 2005 Jun;50(6):725-39; discussion 739-41. PMID 15913465
- [Result] Shorr AF, Kollef MH. Ventilator-associated pneumonia: insights from recent clinical trials. Chest. 2005 Nov;128(5 Suppl 2):583S-591S. doi: 10.1378/chest.128.5_suppl_2.583S. PMID 16306057
- [Result] Thompson DA, Makary MA, Dorman T, Pronovost PJ. Clinical and economic outcomes of hospital acquired pneumonia in intra-abdominal surgery patients. Ann Surg. 2006 Apr;243(4):547-52. doi: 10.1097/01.sla.0000207097.38963.3b. PMID 16552208
- [Result] Yoon, M. & Steele, C. The oral care imperative: The link between oral hygiene and aspiration pneumonia. Topics in Geriatric Rehabilitation. 23(3), 280-288.
- [Result] Shi Z, Xie H, Wang P, Zhang Q, Wu Y, Chen E, Ng L, Worthington HV, Needleman I, Furness S. Oral hygiene care for critically ill patients to prevent ventilator-associated pneumonia. Cochrane Database Syst Rev. 2013 Aug 13;(8):CD008367. doi: 10.1002/14651858.CD008367.pub2. PMID 23939759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The retrospective study group included care-dependent adults with a primary diagnosis of neurological injury/insult (n=51) meeting the inclusion criteria. Enrolled subjects in the prospective study received the experimental protocol (n=32).
Groups:
- Retrospective Study Group: A retrospective chart review identified matched in-patients meeting the study inclusion criteria.
- Oral Care Treatment Group: All subjects in the intervention group received the enhanced oral care protocol:
  * Changing mouth suction equipment every 24 hours
  * Mouth assessment every 2-4 hours
  * Cleansing mouth with toothbrush every 12 hours
  * Cleansing oral mucosa with oral rinse solution every 2-4 hours
  * Moisturize mouth/lips with swab and standard mouth moisturizer every 4 hours
  * Suction mouth and throat as needed
  * Head of the bed elevated to a minimum of 30° during oral care
Period: Overall Study
Arm/Group | Retrospective Study Group | Oral Care Treatment Group
Started | 51 | 32
Completed | 51 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oral Care Treatment Group: Subjects were neurologically impaired, dependent adults who met inclusion criteria. Subjects were identified upon admission to the in-patient unit during the study period.
- Retrospective Study Group: Subjects were neurologically impaired, dependent adults who met inclusion criteria. Subjects were identified through a retrospective chart review for the same in-patient unit.
- Total: Total of all reporting groups
Arm/Group | Oral Care Treatment Group | Retrospective Study Group | Total
Number analyzed (Participants) | 32 | 51 | 83
Age, Customized [Number; unit: participants]
  Age >=19 | 32 | 51 | 83
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 24 | 33
  Male | 23 | 27 | 50
Region of Enrollment [Number; unit: participants] — The study was conducted on a 31 bed acute neurosurgical unit at a tertiary care trauma hospital in Western Canada. The hospital is one of 12 acute care centers in a large metropolitan health region. The study unit was outside of critical care environments. Unit staff consists of a mix of novice and experienced staff including registered nurses (RNs), licensed practice nurses (LPNs), patient care assistants (PCAs), and a rehabilitation team.
  participants
    Canada | 32 | 51 | 83

OUTCOME MEASURES:

1. Primary Outcome: Hospital Acquired Pneumonia Occurrences
Description: Hospital acquired pneumonia is acquired greater than 48 hours after admission and is diagnosed by a positive chest x-ray plus 2 of the following 3 symptoms: presence of fever, elevated serum white blood cells count, and positive sputum specimen.
Time Frame: 10 months
Measure: Number; unit: participants
Groups:
- Oral Care Treatment Group: Acute neurologically impaired adults receiving the study protocol
- Retrospective Study Group: Acute neurologically impaired adults in the retrospective chart review
Arm/Group | Oral Care Treatment Group | Retrospective Study Group
Number analyzed (Participants) | 32 | 51
participants | 2 | 13

ADVERSE EVENTS:
Time Frame: 6 months.
Description: Participants experience included total time receiving treatment up to and not exceeding 6 months.
Groups:
- Oral Care Treatment Group: Subjects meeting the inclusion criteria and identified at the point of admission to the in-patient unit during the study period.
- Retrospective Study Group: Subjects were identified through a chart review process for in-patients on the study unit unit during the retrospective study period and met the inclusion criteria .
Arm/Group | Oral Care Treatment Group | Retrospective Study Group
Serious Adverse Events (participants affected / at risk) | 2/32 | 13/51
Other Adverse Events (participants affected / at risk) | 0/32 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Care Treatment Group (N=32) | Retrospective Study Group (N=51)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 13 (13) — 2/32 study subjects acquired pneumonia while on the protocol

LIMITATIONS AND CAVEATS:
This study was supported by the Fraser Health Point of Care Research Challenge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes